CLINICAL TRIAL: NCT06612957
Title: A Randomized Controlled Study of Uterine Incision Diverticular Repair During Repeated Cesarean Section
Brief Title: A Randomized Controlled Study of Uterine Incision Diverticulum Repair vs. no Repair During Second/Third Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai First Maternal and Infant Health Hospital affiliated to Tongji University Medical School (Other)
Responsible Party: Principal Investigator, Xiaohua Liu, senior chief physician, Shanghai First Maternal and Infant Health Hospital affiliated to Tongji University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024B06
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cesarean Scar Diverticulum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cesarean Section + Uterine Diverticulum Repair Group (Experimental): The original skin incision is used as the surgical incision. Tissues are sequentially separated until reaching the uterus. The original uterine incision'supper edge is used as the surgical incision for this procedure. The bladder is pushed down to fully expose the lower segment of the uterus. After the complete delivery of the fetus and placenta, the placental tissues are thoroughly cleaned, and the uterine scar diverticulum tissue in the lower segment is trimmed down to the original incision edge, making the lower edge of the incision normal uterine muscle tissue. The trimmed uterine scar diverticulum tissue is sent for pathological examination.
  Interventions: Procedure: Repair of uterine cicatricial diverticulum
- Conventional Surgery Group (No Intervention): Participants randomly assigned to the control group undergo the same preoperative preparations and surgical procedures as the intervention group, except for the specific steps involving the repair of the uterine diverticulum.

INTERVENTIONS:
Procedure: Repair of uterine cicatricial diverticulum — Cut off the uterine cicatricial diverticular tissue in the lower portion of the uterus, and restore normal uterine muscle tissue.
  Arms: Cesarean Section + Uterine Diverticulum Repair Group

SUMMARY:
The goal of this study is to assess the efficacy and safety of uterine incision diverticulum repair during repeat cesarean section.The main questions it aims to answer are:

* Can this surgical method improve the symptom of menorrhagia？
* Is this procedure safe？ Researchers will compare experimental group(Cesarean section + diverticulum repair group) to control group(Conventional cesarean section group) to see if this surgical method works to treat or improve menorrhagia.

Participants will:

* randomly assigned 1:1 to the experimental group（repairing uterine diverticula during cesarean section) and the control group （Routine cesarean section without repairing the uterine incision diverticulum）
* visit the hospital 42 days after surgery
* followed up by telephone 6-12 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years, gestational age ≥37 weeks, singleton pregnancy, previous lower segment cesarean section, second or third cesarean section, and diagnosed with uterine incision diverticulum by imaging before or during early pregnancy.

Exclusion Criteria:

* Preoperative indications of placenta accreta or previa, interdelivery interval less than 18 months from the last cesarean section, history of other uterine surgeries, and severe obstetric or medical complications requiring emergency care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Regularity of postpartum menstrual cycle | Six months after cesarean section
  Whether the symptoms of menorrhagia after cesarean section disappear or improve

IPD SHARING:
Plan to Share IPD: No
no share